CLINICAL TRIAL: NCT02723786
Title: A Phase 2 Pilot, Multicenter, Single Arm Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of GSK1070806 Plus Standard of Care for the Prevention of Delayed Graft Function in Adult Subjects After Renal Transplantation
Brief Title: Efficacy, Safety, Tolerability and Pharmacokinetic (PK) Study of GSK1070806 for the Prevention of Delayed Graft Function (DGF) in Adult Subjects After Renal Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 204824; 2015-002812-33 (EudraCT Number)
Record Dates: First submitted 2016-03-14; First posted 2016-03-30 (Estimated); Results first posted 2019-06-10 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-05

CONDITIONS: Kidney Transplantation (Status Post)
Keywords: Delayed Graft Function; Renal Transplantation; Prevention; GSK1070806
MeSH Terms: conditions — Delayed Graft Function | interventions — GSK1070806; Mycophenolic Acid; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GSK1070806 3 mg/kg IV (Experimental): Subjects received a single dose of 3 milligram per kilogram (mg/kg) intravenous (IV) infusion of GSK1070806 administered prior to kidney allograft reperfusion. Subjects also received a combination immunosuppression comprized of basiliximab; mycophenolate mofetil (MMF) or aziothioprine; tacrolimus; and corticosteroids based on the clinical judgment of the investigator.
  Interventions: Biological: GSK1070806; Drug: 1) basiliximab 2) mycophenolate mofetil (MMF) OR azathioprine 3) tacrolimus 4) corticosteroids

INTERVENTIONS:
Biological: GSK1070806 — Injectable solution of 100 milligram/millilitre (mg/mL), administered as a single dose of 3 milligram/kilogram (mg/kg) (maximum of 10 mg/kg) diluted in 100 mL sterile IV infusion bag of 0.9% Sodium Chloride.
Drug: 1) basiliximab 2) mycophenolate mofetil (MMF) OR azathioprine 3) tacrolimus 4) corticosteroids — This immunosuppressant regimen may be revised based on the clinical judgment of the investigator including titration of tacrolimus levels.

SUMMARY:
This is a phase 2 study to evaluate the efficacy, safety, tolerability and pharmacokinetics of GSK1070806 in subjects undergoing renal transplantation. GSK1070806 is an anti-interleukin 18 (IL18) monoclonal antibody, which binds to IL-18 and inhibits signaling through the IL-18 receptor. Recipients of donor kidneys, retrieved after circulatory death of the donor, will be administered a single intravenous infusion of GSK1070806 to test whether inhibition of IL-18 can reduce the rate of Delayed Graft Function (DGF) and graft rejection. Subjects will be followed for 12 months post dose/transplant. Up to 40 adult subjects will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Recipient age range: Between 18 and 75 years of age inclusive, at the time of signing the informed consent.
* Dialysis-dependent recipient of first time, single kidney-only, Donation after Circulatory Death (DCD) transplant.
* Eligible for kidney transplantation: Considered eligible after undergoing multidisciplinary evaluation at the institution at which the transplantation will be performed.
* Immunosuppressants (at the time of transplantation): planned to receive a combination of immunosuppressants including basiliximab, mycophenolate mofetil or azathioprine, tacrolimus, and corticosteroids.
* Male and Female:

  1. Males: Male subjects with female partners of child bearing potential must utilize a condom and female partners must comply with use of highly effective contraceptive methods for 180 days post-dose of study medication.
  2. Females:

     * Non-reproductive potential defined as in the protocol. Reproductive potential: Must not be pregnant or lactating, and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) for 180 days post dose as defined in the protocol.
* Capable of providing signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in the protocol.

Exclusion Criteria:

* Liver function: Alanine Aminotransferase (ALT) >2xUpper Limit of Normal (ULN) and bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* QT interval: single or average Corrected QT Interval (QTc)>480 milliseconds (msec) or in subjects with bundle branch block QTc>500 msec (these criteria do not apply to subjects with predominately paced rhythms).
* Concurrent medication: Subjects who receive treatment that is prohibited for safety reasons (e.g. live vaccines, cyclophosphamide or other biologic immunosuppressants) should not receive investigational product without the explicit approval of the Medical Monitor (Sponsor).
* Investigational product: Any within 5 half-lives or twice the duration of the biological effect whichever is longer (investigational product refers to any drug not approved for sale in the country in which it is being used).
* Immunosuppression: Are being considered for steroid-free, anti-thymocyte globulin (ATG) or alemtuzumab induction, which have a much more profound and prolonged immunosuppressive effect than basiliximab.
* Prior biologic immunosuppressives: The subject has received an agent within the following time period prior to the day of dosing in the current study: 30 days, 5 half-lives or twice the duration of the biological effect, whichever is longer.
* Vaccines: A live vaccine within 30 days prior to GSK1070806 administration
* Receiving a DCD kidney allograft from a donor with any of the following characteristics: cold ischemic time >36 hours, age <5 years old, age >75 years old, ABO blood type incompatible against the recipient, T- and/or B-cell positive cross-match by complement dependent cytotoxicity or flow cytometry against the recipient (where positive cross-match is unavailable, virtual cross-match is allowed), serology positive for hepatitis B (except hepatitis B surface antibody and prior vaccination), hepatitis C or human immunodeficiency virus (HIV), Epstein Barr Virus (EBV) positive donor allograft with an EBV negative recipient, donor had acute or chronic bacterial, viral or fungal infection that according to the investigator causes a risk to recipient, particularly if the infection was resistant or systemic, normothermic regional machine perfusion organ retrieval techniques were utilized, surgical damage to donor allograft during organ procurement
* Previous organ transplantation: has previously undergone any other organ transplantation (with the exception of corneal transplantation).
* Malignancy: has a history of malignancy in the past 5 years except for adequately treated cancers of the skin (basal or squamous cell) or carcinoma in situ of the uterine cervix.
* Acute or chronic infection: has required management of acute or chronic infections (excludes prophylaxis of infections), as follows: currently being treated for a chronic infection, which in the opinion of the investigator, could put the subject at undue risk; hospitalized for treatment of infection, or treated for an infection with parenteral antibiotics (includes antibacterials, antivirals, anti-fungals, or anti-parasitic agents) within 30 days before Day 0, which in the opinion of the investigator, could put the subject at undue risk; current evidence, or history within the last 14 days, of an influenza-like illness as defined by fever (>38 degree Celsius) and two or more of the following symptoms: cough, sore throat, runny nose, sneezing, limb / joint pain, headache, vomiting / diarrhoea; subjects with any history of active tuberculosis, recent tuberculosis exposure, or judged by investigators to be at risk of tuberculosis will be excluded from the study.
* Other disease/conditions. Has any of the following: clinical evidence of significant unstable or uncontrolled acute or chronic diseases, which in the opinion of the investigator, could confound the results of the study or put the subject at undue risk; a surgical procedure planned in the 12 months after Day 0, other than kidney transplantation or related procedure; a known history of any other medical disease (e.g., cardiopulmonary), laboratory abnormality, or condition (e.g., poor venous access) that, in the opinion of the investigator, makes the subject unsuitable for the study
* Hepatitis B: subjects will be excluded with any evidence of acute or chronic infection, or if interpretation of their results is unclear. This includes: Hepatitis B surface Antigen (HBsAg)+, Anti- Hepatitis B core (Anti-HBc)+, Hepatitis B Deoxyribose Nucleic Acid (HB DNA)+. It is permissible to enroll subjects who are anti-Hepatitis B (HB)s+ only, when this is attributable to vaccination and there is no history of previous infection.
* Hepatitis C: subjects will be excluded if there is any evidence of past or current hepatitis C infection, including hepatitis C antibody, hepatitis C Recombinant ImmunoBlot Assay (RIBA) or Polymerase Chain Reaction (PCR).
* HIV: known to have a historically positive HIV test.
* Immunodeficiency: recipient with a history of, or laboratory evidence of immunodeficiency.
* Drug Sensitivity: has a history of sensitivity to any of the study medications including: GSK1070806; background immunosuppressive regimen; designated prophylactic anti-infective therapies or components thereof, or a history of drug or other allergy including a previous anaphylactic reaction to parenteral administration or biologic therapy (ie monoclonal antibody) that, in the opinion of the Investigator or Medical Monitor, contraindicates their participation.
* Substance abuse: has clinical evidence of current drug or alcohol abuse or dependence.
* Co enrollment: participating in another interventional study (participation in purely observational or cohort studies is acceptable provided they do not impair feasibility, or involve excessive additional sampling).
* Compliance: is unlikely to comply with scheduled study visits based on investigator judgment or has a history of a psychiatric disorder or condition that may compromise communication with the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-08-27 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2018-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- GSK Investigational Site, L'Hospitalet de Llobregat, Spain
- United Kingdom (3):
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Wlodek E, Kirkpatrick RB, Andrews S, Noble R, Schroyer R, Scott J, Watson CJE, Clatworthy M, Harrison EM, Wigmore SJ, Stevenson K, Kingsmore D, Sheerin NS, Bestard O, Stirnadel-Farrant HA, Abberley L, Busz M, DeWall S, Birchler M, Krull D, Thorneloe KS, Weber A, Devey L. A pilot study evaluating GSK1070806 inhibition of interleukin-18 in renal transplant delayed graft function. PLoS One. 2021 Mar 8;16(3):e0247972. doi: 10.1371/journal.pone.0247972. eCollection 2021. PMID 33684160

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single arm study to evaluate the efficacy, safety, tolerability, and pharmacokinetics (PK) of GSK1070806 plus standard of care (SOC) for the prevention of delayed graft function in adult participants after renal transplantation.
Pre-assignment Details: A total of 10 participants were screened for the study, and 7 of them received study treatment. The study enrolled participants in 4 centers across 2 countries (Spain and United Kingdom).
Groups:
- GSK1070806 3 mg/kg IV: Participants received a single dose of 3 milligram per kilogram (mg/kg) intravenous (IV) infusion of GSK1070806 administered prior to kidney allograft reperfusion. Participants also received a combination immunosuppression comprised of basiliximab; mycophenolate mofetil (MMF) or aziothioprine; tacrolimus; and corticosteroids based on the clinical judgment of the investigator.
Period: Overall Study
Arm/Group | GSK1070806 3 mg/kg IV
Started | 7
Completed | 6
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | GSK1070806 3 mg/kg IV
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.7 (13.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Requiring Dialysis During the First 7 Days Post Transplant
Description: The requirement of dialysis (except as needed for hyperkalaemia during the first 24 hours [hrs]) were used to assess the frequency of delayed graft function (DGF) in donation after circulatory death (DCD) renal transplant recipients treated with GSK1070806. The 'Analysis Population' (AP) is defined as participants in the 'All Subjects' Population who have been declared to have DGF or have reached 7 days.
Time Frame: Up to Day 7
Population: AP Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1070806 3 mg/kg IV
Number analyzed (Participants) | 7
Participants | 4
Statistical Analysis 1: Comparison: GSK1070806 3 mg/kg IV; Test type: Other; The proportion of participants with DGF was 0.57, highest Posterior Density (HPD) 95% Credible interval (CI) (0.25,0.90). The posterior probability for the proportion of participants with DGF <30% was 0.07 (HPD 95% CI [0.00,1.00]). The posterior probability for the proportion of participants with DGF <50% was 0.34 (HPD 95% CI [0.00,1.00])

2. Secondary Outcome: Serum Creatinine at Baseline and Change From Baseline Over Time Post Transplant
Description: Blood samples were collected to measure serum creatinine at the indicated timepoints to assess graft function in DCD renal transplant recipients treated with GSK1070806. Baseline value was the latest pre-dose assessment value. Change from Baseline was post Baseline value minus Baseline value. NA indicates data is not available as standard deviation could not be calculated due to n=1. The AP Population is defined as participants having Baseline and at least one post-Baseline assessment.
Time Frame: Baseline and up to 12 months
Population: AP Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | GSK1070806 3 mg/kg IV
Number analyzed (Participants) | 7
Micromoles per liter
  Screening, n=7 | 679.0 (175.14)
  Day 0, n=7 | -39.3 (160.09)
  Day 1, n=7 | -44.7 (214.06)
  Day 2, n=7 | -99.0 (304.29)
  Day 3, n=7 | -36.7 (378.28)
  Day 4, n=7 | -104.6 (378.79)
  Day 5, n=6: number analyzed (Participants) | 6
  Day 5, n=6 | -57.2 (334.19)
  Day 6, n=6: number analyzed (Participants) | 6
  Day 6, n=6 | -75.7 (308.22)
  Day 7, n=6: number analyzed (Participants) | 6
  Day 7, n=6 | -43.5 (321.91)
  Day 8, n=5: number analyzed (Participants) | 5
  Day 8, n=5 | -150.8 (293.48)
  Day 9, n=3: number analyzed (Participants) | 3
  Day 9, n=3 | -24.0 (297.82)
  Day 10, n=3: number analyzed (Participants) | 3
  Day 10, n=3 | -53.0 (395.94)
  Day 11, n=3: number analyzed (Participants) | 3
  Day 11, n=3 | -97.0 (462.46)
  Day 12, n=2: number analyzed (Participants) | 2
  Day 12, n=2 | 110.0 (257.39)
  Day 13, n=2: number analyzed (Participants) | 2
  Day 13, n=2 | 38.0 (209.30)
  Day 14, n=2: number analyzed (Participants) | 2
  Day 14, n=2 | 4.0 (190.92)
  Day 15, n=2: number analyzed (Participants) | 2
  Day 15, n=2 | -51.0 (172.53)
  Day 16, n=2: number analyzed (Participants) | 2
  Day 16, n=2 | -61.5 (173.24)
  Day 17, n=2: number analyzed (Participants) | 2
  Day 17, n=2 | -107.5 (143.54)
  Day 18, n=2: number analyzed (Participants) | 2
  Day 18, n=2 | -145.0 (123.04)
  Day 19, n=2: number analyzed (Participants) | 2
  Day 19, n=2 | -173.5 (95.46)
  Day 20, n=2: number analyzed (Participants) | 2
  Day 20, n=2 | -183.5 (81.32)
  Day 21, n=1: number analyzed (Participants) | 1
  Day 21, n=1 | -117.0 (NA) — Standard deviation could not be calculated due to n=1.
  Day 22, n=1: number analyzed (Participants) | 1
  Day 22, n=1 | -91.0 (NA) — Standard deviation could not be calculated due to n=1.
  Day 23, n=1: number analyzed (Participants) | 1
  Day 23, n=1 | -95.0 (NA) — Standard deviation could not be calculated due to n=1.
  Day 24, n=1: number analyzed (Participants) | 1
  Day 24, n=1 | -115.0 (NA) — Standard deviation could not be calculated due to n=1.
  Day 25, n=1: number analyzed (Participants) | 1
  Day 25, n=1 | -152.0 (NA) — Standard deviation could not be calculated due to n=1.
  Day 26, n=1: number analyzed (Participants) | 1
  Day 26, n=1 | -155.0 (NA) — Standard deviation could not be calculated due to n=1.
  Day 27, n=1: number analyzed (Participants) | 1
  Day 27, n=1 | -175.0 (NA) — Standard deviation could not be calculated due to n=1.
  Day 28, n=1: number analyzed (Participants) | 1
  Day 28, n=1 | -191.0 (NA) — Standard deviation could not be calculated due to n=1.
  Day 30, n=7 | -478.3 (225.47)
  Day 90, n=7 | -489.9 (214.06)
  6 months, n=7 | -467.4 (232.49)
  12 months, n=6: number analyzed (Participants) | 6
  12 months, n=6 | -490.5 (224.32)

3. Secondary Outcome: Urine Volume at Baseline and Change From Baseline Over Time Post Transplant
Description: Urine volume at Baseline and over time post transplant was measured to assess graft function in DCD renal transplant recipients treated with GSK1070806. Baseline value was the latest pre-dose assessment value. Change from Baseline was post Baseline value minus Baseline value. All Subjects Population comprised of participants who received the dose of study medication.
Time Frame: Baseline (Pre-operative) and up to Day 28
Population: All Subjects Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | GSK1070806 3 mg/kg IV
Number analyzed (Participants) | 7
Liter
  Baseline (Pre-operative), n=5: number analyzed (Participants) | 5
  Baseline (Pre-operative), n=5 | 0.6700 (0.60581)
  Day 0, n=4: number analyzed (Participants) | 4
  Day 0, n=4 | -0.5150 (0.59533)
  Day 1, n=5: number analyzed (Participants) | 5
  Day 1, n=5 | 0.5862 (1.56917)
  Day 2, n=5: number analyzed (Participants) | 5
  Day 2, n=5 | 1.2820 (2.62989)
  Day 3, n=5: number analyzed (Participants) | 5
  Day 3, n=5 | 0.8840 (1.04040)
  Day 4, n=5: number analyzed (Participants) | 5
  Day 4, n=5 | 1.1480 (1.00442)
  Day 5, n=4: number analyzed (Participants) | 4
  Day 5, n=4 | 0.8270 (1.02297)
  Day 6, n=4: number analyzed (Participants) | 4
  Day 6, n=4 | 1.1168 (1.30252)
  Day 7, n=4: number analyzed (Participants) | 4
  Day 7, n=4 | 1.2985 (1.37212)
  Day 8, n=3: number analyzed (Participants) | 3
  Day 8, n=3 | 1.2090 (1.20354)
  Day 9, n=2: number analyzed (Participants) | 2
  Day 9, n=2 | 1.2135 (1.46866)
  Day 10, n=2: number analyzed (Participants) | 2
  Day 10, n=2 | 0.8585 (0.62720)
  Day 11, n=2: number analyzed (Participants) | 2
  Day 11, n=2 | 0.4985 (0.22840)
  Day 12, n=1: number analyzed (Participants) | 1
  Day 12, n=1 | 1.4000 (NA) — Standard deviation could not be calculated due to n=1.
  Day 13, n=1: number analyzed (Participants) | 1
  Day 13, n=1 | 1.6900 (NA) — Standard deviation could not be calculated due to n=1.
  Day 14, n=1: number analyzed (Participants) | 1
  Day 14, n=1 | 1.1800 (NA) — Standard deviation could not be calculated due to n=1.
  Day 15, n=1: number analyzed (Participants) | 1
  Day 15, n=1 | 1.5500 (NA) — Standard deviation could not be calculated due to n=1.
  Day 16, n=1: number analyzed (Participants) | 1
  Day 16, n=1 | 1.8500 (NA) — Standard deviation could not be calculated due to n=1.
  Day 17, n=1: number analyzed (Participants) | 1
  Day 17, n=1 | 1.5000 (NA) — Standard deviation could not be calculated due to n=1.
  Day 18, n=1: number analyzed (Participants) | 1
  Day 18, n=1 | 1.9000 (NA) — Standard deviation could not be calculated due to n=1.
  Day 19, n=1: number analyzed (Participants) | 1
  Day 19, n=1 | 1.6000 (NA) — Standard deviation could not be calculated due to n=1.
  Day 20, n=1: number analyzed (Participants) | 1
  Day 20, n=1 | 1.2500 (NA) — Standard deviation could not be calculated due to n=1.
  Day 21, n=1: number analyzed (Participants) | 1
  Day 21, n=1 | 0.7500 (NA) — Standard deviation could not be calculated due to n=1.
  Day 22, n=1: number analyzed (Participants) | 1
  Day 22, n=1 | 1.0500 (NA) — Standard deviation could not be calculated due to n=1.
  Day 23, n=1: number analyzed (Participants) | 1
  Day 23, n=1 | 1.1500 (NA) — Standard deviation could not be calculated due to n=1.
  Day 24, n=1: number analyzed (Participants) | 1
  Day 24, n=1 | 1.4500 (NA) — Standard deviation could not be calculated due to n=1.
  Day 25, n=1: number analyzed (Participants) | 1
  Day 25, n=1 | 2.0500 (NA) — Standard deviation could not be calculated due to n=1.
  Day 26, n=1: number analyzed (Participants) | 1
  Day 26, n=1 | 2.0000 (NA) — Standard deviation could not be calculated due to n=1.
  Day 27, n=1: number analyzed (Participants) | 1
  Day 27, n=1 | 1.5500 (NA) — Standard deviation could not be calculated due to n=1.
  Day 28, n=1: number analyzed (Participants) | 1
  Day 28, n=1 | 1.4600 (NA) — Standard deviation could not be calculated due to n=1.

4. Secondary Outcome: Number of Participants in the First 7 Days With: Primary Non Function, Functional DGF, Intermediate Graft Function, Immediate Graft Function
Description: Number of participants in the first 7 days with primary non function, functional DGF, intermediate graft function and immediate graft function were evaluated to access graft function in DCD renal transplant recipients treated with GSK1070806. The AP Population is defined as participants in the 'All Subjects' Population who have been declared to have DGF or have reached 7 days.
Time Frame: Up to Day 7
Population: All Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1070806 3 mg/kg IV
Number analyzed (Participants) | 7
Participants
  Primary Non Function | 1
  3 day Functional DGF | 3
  7 day Functional DGF | 5
  3 day Intermediate Graft Function | 0
  7 day Intermediate Graft Function | 1
  3 day Immediate Graft Function | 1
  7 day Immediate Graft Function | 0

5. Secondary Outcome: Number of Participants With Episodes of Biopsy-proven Acute Rejection
Description: Number of participants with episodes of biopsy-proven acute rejection were evaluated to assess the effect of GSK1070806 on acute rejection risk, and rejection/Pharmacodynamic (PD) biomarkers.
Time Frame: Up to 12 months
Population: All Subjects Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1070806 3 mg/kg IV
Number analyzed (Participants) | 2
Participants | 1

6. Secondary Outcome: Serum Interferon Gamma-induced Protein 10 (IP-10) and Serum Monokine Induced Gamma Interferon (Mig) Levels at Baseline and Change From Baseline Over Time Post Transplant
Description: The interferon-gamma -inducible chemokine IP10 and the interferon-gamma -inducible chemokine Mig have been identified as an early predictive marker of antibody-mediated kidney graft rejection. Baseline value was the latest pre-dose assessment value. Change from Baseline was calculated as post Baseline value minus Baseline value.
Time Frame: Baseline and at 0.75 hours, 4-8 hours, Day 1, Day 2, Day 30, Day 90, 6 months and 12 months post reperfusion
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Picograms per milliliter
Arm/Group | GSK1070806 3 mg/kg IV
Number analyzed (Participants) | 7
Picograms per milliliter
  IP-10, Baseline, n=7 | 518.83817 (269.010355)
  IP-10, Day 0, 0.75 hour, n=6: number analyzed (Participants) | 6
  IP-10, Day 0, 0.75 hour, n=6 | -48.36607 (178.371827)
  IP-10, Day 0, 4-8 hour, n=6: number analyzed (Participants) | 6
  IP-10, Day 0, 4-8 hour, n=6 | -262.30099 (176.415675)
  IP-10, Day 1, n=6: number analyzed (Participants) | 6
  IP-10, Day 1, n=6 | -214.27224 (198.587957)
  IP-10, Day 2, n=5: number analyzed (Participants) | 5
  IP-10, Day 2, n=5 | -91.07498 (397.795706)
  IP-10, Day 30, n=6: number analyzed (Participants) | 6
  IP-10, Day 30, n=6 | -215.96831 (350.419207)
  IP-10, Day 90, n=7 | 221.97286 (617.906913)
  IP-10, 6 months, n=7 | 145.05039 (846.080946)
  IP-10, 12 months, n=5: number analyzed (Participants) | 5
  IP-10, 12 months, n=5 | 241.29317 (564.374462)
  Mig, Baseline, n=7 | 175.76865 (194.372235)
  Mig, Day 0, 0.75 hour, n=6: number analyzed (Participants) | 6
  Mig, Day 0, 0.75 hour, n=6 | -14.02145 (32.535124)
  Mig, Day 0, 4-8 hour, n=6: number analyzed (Participants) | 6
  Mig, Day 0, 4-8 hour, n=6 | -49.28436 (54.067623)
  Mig, Day 1, n=6: number analyzed (Participants) | 6
  Mig, Day 1, n=6 | -67.61716 (61.009544)
  Mig, Day 2, n=5: number analyzed (Participants) | 5
  Mig, Day 2, n=5 | -133.99600 (165.972042)
  Mig, Day 30, n=6: number analyzed (Participants) | 6
  Mig, Day 30, n=6 | -159.17646 (207.921389)
  Mig, Day 90, n=7 | -78.69081 (227.901113)
  Mig, 6 months, n=7 | -43.68148 (325.518838)
  Mig, 12 months, n=5: number analyzed (Participants) | 5
  Mig, 12 months, n=5 | -30.52711 (75.218188)

7. Secondary Outcome: Number of Participants With Dialysis Events in the First 30 Days Post-transplant
Description: Number of participants with dialysis events in the first 30 days post transplant was evaluated to assess the effect of GSK1070806 on dialysis dependency and graft survival. The AP Population is defined as participants having Baseline and at least one post-Baseline assessment.
Time Frame: Up to 30 days
Population: AP Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1070806 3 mg/kg IV
Number analyzed (Participants) | 7
Participants | 5

8. Secondary Outcome: Number of Participants Who Are Dialysis Independent at Visits up to 12 Months Post-transplant
Description: Number of participants who are dialysis independent at visits up to 12 months post transplant was evaluated to assess the effect of GSK1070806 on dialysis dependency and graft survival.
Time Frame: Up to 12 months
Population: All Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1070806 3 mg/kg IV
Number analyzed (Participants) | 7
Participants | 2

9. Secondary Outcome: Number of Participants With Adverse Event (AE) and Serious Adverse Event (SAE)
Description: AE is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment were categorized as SAE.
Time Frame: Up to 12 months
Population: All Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1070806 3 mg/kg IV
Number analyzed (Participants) | 7
Participants
  Any AE | 7
  Any SAE | 6

10. Secondary Outcome: Number of Participants Having Any Abnormality in Hematology Results of Potential Clinical Importance
Description: Blood samples were collected to evaluate hematology parameters. Number of participants with abnormality in any hematology parameter results of potential clinical importance (high or low) observed at any time post Baseline are presented. PCI (high or low) was considered if hematocrit (high:>0.54;low:change from baseline [CFB] 0.075 decrease), hemoglobin (high:180; low: CFB 25 decrease), lymphocytes (low: 0.8), neutrophil count (low: 1.5), platelet count (low: 100; high: 550), White blood cells (low: 3; high:20).
Time Frame: Up to 12 months
Population: All Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1070806 3 mg/kg IV
Number analyzed (Participants) | 7
Participants
  Lymphocytes, Low | 7
  Hematocrit, High | 1
  White Blood Cells, High | 1
  White Blood Cells, Low | 1
  Platelet Count, Low | 1
  Total neutrophils, Low | 1

11. Secondary Outcome: Number of Participants Having Any Abnormal Clinical Chemistry Results of Potential Clinical Importance
Description: Blood samples were collected to evaluate clinical chemistry parameters. Number of participants with abnormal chemistry results of potential clinical importance (high or low) in any of these parameters at any time post Baseline visit have been presented. PCI (high or low) was considered if albumin (low<30), calcium (low<2, high>2.75), creatinine (high: CHB>44.2 increase), glucose (low<3, high>9), magnesium (low<0.5, high>1.23), phosphorus (low<0.8, high>1.6), potassium (low<3, high>5.5), sodium (low: 130, high>150), Total carbon dioxide (CO2) (low:18, high>32), Alanine aminotransferase (ALT) (high>=2*upper limit of normal [ULN]), Aspartate aminotransferase (AST) (high: >=2*ULN), Alkaline phosphatase (ALP) (high:>=2*ULN), Total bilirubin (high: >2*ULN), Total bilirubin+ALT (high: 1.5*ULN total bilirubin with >=2*ULN ALT).
Time Frame: Up to 12 months
Population: All Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1070806 3 mg/kg IV
Number analyzed (Participants) | 7
Participants
  Albumin, Low | 6
  Calcium, Low | 7
  Glucose, High | 5
  Potassium, Low | 1
  Potassium, High | 3
  Total Bilirubin, High | 1
  Sodium, Low | 2
  ALT, High | 1
  ALP, High | 1
  AST, High | 1

12. Secondary Outcome: Number of Participants Having Any Abnormality of Potential Clinical Importance of Vital Signs Results
Description: Vital signs parameters included analysis of systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate (HR) and body temperature. Number of participants with any abnormality of potential clinical importance (high or low) in any of these vitals signs at any time post Baseline visit have been presented. PCI (high or low) was considered if SBP (low: <85, high:>160), DBP (low: <45, high>100), HR (low: <40, high: >110) and temperature (low: <35.5, high: >37.5).
Time Frame: Up to 12 months
Population: All Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1070806 3 mg/kg IV
Number analyzed (Participants) | 7
Participants
  SBP, High | 5
  SBP, Low | 1
  DBP, High | 2
  DBP, Low | 1
  HR, High | 1
  Temperature, High | 1
  Temperature, Low | 2

13. Secondary Outcome: Number of Participants Having Infections
Description: Number of participants having infections were summarized.
Time Frame: Up to 12 months
Population: All Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1070806 3 mg/kg IV
Number analyzed (Participants) | 7
Participants | 5

14. Secondary Outcome: Serum Concentrations of GSK1070806
Description: Serial blood samples were collected to evaluate PK of GSK1070806 at Pre-operative, 0.75 hours, 4-8 hours, 24 hours, 168 hours, Day 30, Day 90, 6 months and 12 months after kidney reperfusion. PK Population included participants in the 'All Subjects' Population for whom a serum PK sample is obtained and analyzed for GSK1070806.
Time Frame: Pre-operative, 0.75 hours, 4-8 hours, 24 hours, 168 hours, Day 30, Day 90, 6 months and 12 months after kidney reperfusion
Population: PK Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | GSK1070806 3 mg/kg IV
Number analyzed (Participants) | 7
Nanograms per milliliter
  Pre-operative, n=7 | 0.0 (NA) — Standard deviation is not calculated as most of the values at this time point were imputed.
  0.75 hours, n=6: number analyzed (Participants) | 6
  0.75 hours, n=6 | 58783.3 (11287.77)
  4-8 hours, n=6: number analyzed (Participants) | 6
  4-8 hours, n=6 | 60033.3 (13577.43)
  24 hours, n=6: number analyzed (Participants) | 6
  24 hours, n=6 | 50933.3 (12681.11)
  168 hours, n=5: number analyzed (Participants) | 5
  168 hours, n=5 | 28260.0 (9643.29)
  Day 30, n=6: number analyzed (Participants) | 6
  Day 30, n=6 | 17366.7 (6809.60)
  Day 90, n=7 | 5047.0 (2914.37)
  6 months, n=7 | 1083.4 (720.18)
  12 months, n=6: number analyzed (Participants) | 6
  12 months, n=6 | 19.2 (NA) — Standard deviation is not calculated as most of the values at this time point were imputed.

15. Secondary Outcome: Maximum Plasma Concentration (Cmax) of GSK1070806
Description: Serial blood samples were collected to evaluate PK of GSK1070806 at Pre-operative, 0.75 hours, 4-8 hours, 24 hours, 168 hours, Day 30, Day 90, 6 months and 12 months after kidney reperfusion. Log-transformed geometric mean and 95% confidence interval have been presented.
Time Frame: as for outcome 14
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: Log (nanograms per milliliter)
Arm/Group | GSK1070806 3 mg/kg IV
Number analyzed (Participants) | 7
Log (nanograms per milliliter) | 36315.1 [10237.6 to 128818.4]

16. Secondary Outcome: Area Under the Plasma Concentration Time Curve (AUC) From Time 0 to the Last Measurable Concentration (AUC[0-t]) and AUC From Time 0 to Infinite Time (AUC[0-inf]) of GSK1070806
Description: Blood samples were collected to evaluate PK of GSK1070806 at Pre-operative, 0.75 hours, 4-8 hours, 24 hours, 168 hours, Day 30, Day 90, 6 months and 12 months after kidney reperfusion. Log-transformed geometric mean and 95% confidence interval have been presented.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Log (Hour*nanograms per milliliter)
Arm/Group | GSK1070806 3 mg/kg IV
Number analyzed (Participants) | 7
Log (Hour*nanograms per milliliter)
  AUC (0-t), n=7 | 26131338.2 [8927844.0 to 76485076.9]
  AUC (0-inf), n=6: number analyzed (Participants) | 6
  AUC (0-inf), n=6 | 41032450.7 [28127219.0 to 59858815.6]

17. Secondary Outcome: Baseline and Change From Baseline in Serum Levels of Free, Total, and GSK1070806 Bound Interleukin 18 (IL-18) Over Time Post-transplant
Description: IL-18 is itself rapidly secreted from intracellular stores following inflammasome mediated-activation. The appearance of IL-18 marks the initiation of the inflammatory response leading to further injury. Blood samples were collected at indicated time points to assess serum levels of free, total, and GSK1070806 bound IL-18. Baseline value was the latest pre-dose assessment value. Change from Baseline was post Baseline value minus Baseline value.
Time Frame: Baseline and at 0.75 hours, 4-8 hours, Day 1, Day 2, Day 30, Day 90, 6 months and 12 months post reperfusion
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Picograms per milliliter
Arm/Group | GSK1070806 3 mg/kg IV
Number analyzed (Participants) | 7
Picograms per milliliter
  Serum Free IL-18, Baseline (pre-operative), n=5: number analyzed (Participants) | 5
  Serum Free IL-18, Baseline (pre-operative), n=5 | 26.840 (37.0569)
  Serum Free IL-18, Day 0, 0.75 hour, n=5: number analyzed (Participants) | 5
  Serum Free IL-18, Day 0, 0.75 hour, n=5 | -22.620 (37.1672)
  Serum Free IL-18, Day 0, 4-8 hour, n=5: number analyzed (Participants) | 5
  Serum Free IL-18, Day 0, 4-8 hour, n=5 | -22.540 (34.1535)
  Serum Free IL-18, Day 1, n=5: number analyzed (Participants) | 5
  Serum Free IL-18, Day 1, n=5 | -23.890 (37.0569)
  Serum Free IL-18, Day 2, n=4: number analyzed (Participants) | 4
  Serum Free IL-18, Day 2, n=4 | -5.263 (14.4846)
  Serum Free IL-18, Day 30, n=4: number analyzed (Participants) | 4
  Serum Free IL-18, Day 30, n=4 | -27.925 (41.5019)
  Serum Free IL-18, Day 90, n=2: number analyzed (Participants) | 2
  Serum Free IL-18, Day 90, n=2 | -2.250 (3.1820)
  Serum Free IL-18, 6 months, n=0: number analyzed (Participants) | 0
  Serum Free IL-18, 12 months, n=0: number analyzed (Participants) | 0
  Serum Bound IL-18, Baseline (pre-operative), n=5: number analyzed (Participants) | 5
  Serum Bound IL-18, Baseline (pre-operative), n=5 | 21.156 (7.5139)
  Serum Bound IL-18, Day 0, 0.75 hour, n=5: number analyzed (Participants) | 5
  Serum Bound IL-18, Day 0, 0.75 hour, n=5 | 362.084 (220.2164)
  Serum Bound IL-18, Day 0, 4-8 hour, n=5: number analyzed (Participants) | 5
  Serum Bound IL-18, Day 0, 4-8 hour, n=5 | 314.864 (139.1919)
  Serum Bound IL-18, Day 1, n=5: number analyzed (Participants) | 5
  Serum Bound IL-18, Day 1, n=5 | 472.204 (193.0366)
  Serum Bound IL-18, Day 2, n=4: number analyzed (Participants) | 4
  Serum Bound IL-18, Day 2, n=4 | 485.740 (252.2876)
  Serum Bound IL-18, Day 30, n=4: number analyzed (Participants) | 4
  Serum Bound IL-18, Day 30, n=4 | 617.543 (282.9679)
  Serum Bound IL-18, Day 90, n=2: number analyzed (Participants) | 2
  Serum Bound IL-18, Day 90, n=2 | 946.020 (21.3971)
  Serum Bound IL-18, 6 months, n=0: number analyzed (Participants) | 0
  Serum Bound IL-18, 12 months, n=0: number analyzed (Participants) | 0
  Serum Total IL-18, Baseline (pre-operative), n=7 | 130.6857 (71.37029)
  Serum Total IL-18, Day 0, 0.75 hour, n=6: number analyzed (Participants) | 6
  Serum Total IL-18, Day 0, 0.75 hour, n=6 | 572.3333 (368.68620)
  Serum Total IL-18, Day 0, 4-8 hour, n=6: number analyzed (Participants) | 6
  Serum Total IL-18, Day 0, 4-8 hour, n=6 | 576.3667 (273.88543)
  Serum Total IL-18, Day 1, n=6: number analyzed (Participants) | 6
  Serum Total IL-18, Day 1, n=6 | 636.5667 (208.88294)
  Serum Total IL-18, Day 2, n=5: number analyzed (Participants) | 5
  Serum Total IL-18, Day 2, n=5 | 660.6600 (297.32305)
  Serum Total IL-18, Day 30, n=6: number analyzed (Participants) | 6
  Serum Total IL-18, Day 30, n=6 | 1175.5000 (710.48323)
  Serum Total IL-18, Day 90, n=7 | 1423.5429 (685.42012)
  Serum Total IL-18, 6 months, n=7 | 1303.7143 (1006.89585)
  Serum Total IL-18, 12 months, n=6: number analyzed (Participants) | 6
  Serum Total IL-18, 12 months, n=6 | 1091.0833 (1102.78861)

18. Secondary Outcome: Number of Participants With Positive Result in Anti-GSK1070806 Antibodies (ADAs)
Description: Serum samples were to be collected to test for the presence of antibodies against GSK1070806 at indicated time points. The presence of anti-GSK1070806 binding antibodies were to be assessed using a validated electrochemiluminescent (ECL) immunoassay.
Time Frame: 0.75 hour and 4-8 hour on Day 0, Day 1, Day 2, Day 30, Day 90, 6 months and 12 months post reperfusion
Population: All Subjects Population. Data was not collected as the immunogenicity samples were not collected for this terminated indication since healthy volunteers showed low titers and Type 2 Diabetics showed no titers per Investigator's Brochure.
Arm/Group | GSK1070806 3 mg/kg IV
Number analyzed (Participants) | 0

19. Secondary Outcome: ADA Titer Before and After GSK1070806 Administration
Description: Serum samples were to be collected to test for the presence of antibodies against GSK1070806 at indicated time points. The presence of ADA titre was to be assessed using a validated ECL immunoassay.
Time Frame: 0.75 hour and 4-8 hour on Day 0, Day 1, Day 2, Day 30, Day 90, 6 months and 12 months post reperfusion
Population: as for outcome 18
Arm/Group | GSK1070806 3 mg/kg IV
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious AEs were defined as events occurring from the first dose until 12 months.
Description: SAEs and Non-serious AEs were collected for All Subjects Population, comprised of participants who received the dose of study medication.
Arm/Group | GSK1070806 3 mg/kg IV
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 6/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1070806 3 mg/kg IV (N=7)
Pneumonia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (3)
Ventricular fibrillation (Cardiac disorders) | 1 (2)
Hernia (General disorders) | 1 (1)
Kidney transplant rejection (Immune system disorders) | 1 (1)
Transplant dysfunction (Injury, poisoning and procedural complications) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ureteral stent removal (Surgical and medical procedures) | 1 (1)
Visceral leishmaniasis (Infections and infestations) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1070806 3 mg/kg IV (N=7)
Constipation (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 5 (5)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (4)
Escherichia urinary tract infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (2)
Postoperative wound infection (Infections and infestations) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (4)
Renal disorder (Renal and urinary disorders) | 1 (1)
Ureteric stenosis (Renal and urinary disorders) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Blood creatine increased (Investigations) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1)
Blood sodium decreased (Investigations) | 1 (1)
Body temperature decreased (Investigations) | 1 (1)
Candida test positive (Investigations) | 1 (1)
Haemoglobin increased (Investigations) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Wound evisceration (Injury, poisoning and procedural complications) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Catheter site haemorrhage (General disorders) | 1 (1)
Kidney transplant rejection (Immune system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Bacterial disease carrier (Infections and infestations) | 1 (1)
Nail infection (Infections and infestations) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 1 (1)
Purulent discharge (Infections and infestations) | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Blood glucose increased (Investigations) | 1 (1)
Cytomegalovirus test positive (Investigations) | 1 (1)
Weight increased (Investigations) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (1)
Post procedural discharge (Injury, poisoning and procedural complications) | 1 (1)
Transplant rejection (Immune system disorders) | 1 (1)
Product contamination (Product Issues) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-05-24): https://cdn.clinicaltrials.gov/large-docs/86/NCT02723786/SAP_000.pdf
  • Study Protocol (2017-05-04): https://cdn.clinicaltrials.gov/large-docs/86/NCT02723786/Prot_001.pdf